CLINICAL TRIAL: NCT06077994
Title: The Enhanced Pulmonary Rehabilitation Program With Digital Remote Patient Monitoring: A Feasibility Randomized Clinical Trial
Brief Title: Enhanced Pulmonary Rehabilitation With Digital Remote Home Monitoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00066560-2
Record Dates: First submitted 2023-09-28; First posted 2023-10-11 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Lung diseases; Pulmonary Rehabilitation; Digital health
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Breathe Easy Pulmonary Rehabilitation Program (BEPR+) (Active Comparator): 6 or 8 weeks BEPR+ program
  Interventions: Behavioral: Enhanced Breathe Easy Pulmonary Rehabilitation Program (BEPR+)
- digital Remote Patient Monitoring + BEPR+ (dRPM+) (Experimental): 6 or 8 weeks BEPR+; daily vitals readings (blood pressure, heart rate, oximetry, body temperature, and body weight) and an additional 12 weeks of dRPM reading once the BEPR+ program concludes
  Interventions: Behavioral: digital Remote Patient Monitoring+BEPR+ (dRPM+)

INTERVENTIONS:
Behavioral: digital Remote Patient Monitoring+BEPR+ (dRPM+) — In addition to the BEPR+ program as described, patients will use the Cloud Dx Connect Health System to take daily physiological readings (Blood pressure, heart rate, oximetry, body temperature and body weight). These data will be transmitted to a secured server supported by the provincial health care system. Participants and therapists will interact with these data in their respective dashboards and in conjunction with participants' determined medical action plan, engage in or make changes to participants current self-management regimens.
  Arms: digital Remote Patient Monitoring + BEPR+ (dRPM+)
Behavioral: Enhanced Breathe Easy Pulmonary Rehabilitation Program (BEPR+) — Patients will attend the BEPR+ program 3 days per week for 6 weeks or 2 days per week for 8 weeks (total of 16 sessions). Patients will receive 90 minutes of personalized and supervised exercise training (aerobic and resistance) and 60 minutes of education designed to promote self-management. Patients will also received one-on-one sessions with a therapist to review their medical action plan for exacerbation management, program and lifestyle goals (including physical activity), determine referral needs for other health services (i.e. smoking cessation, weight management, and psychological support). Patients will use an activity monitor for feedback and motivation for physical activity.
  Arms: Enhanced Breathe Easy Pulmonary Rehabilitation Program (BEPR+)

SUMMARY:
The primary objective of the current randomized controlled trial is to assess feasibility of integrating digital remote patient monitoring (dRPM) with the an enhanced Breathe Easy Pulmonary Rehabilitation Program for Individuals with COPD and Comorbidities (BEPR+), including aspects such as recruitment, retention, patient adherence, technology acceptability, adverse events, and staffing resources. The secondary objectives include comparing clinical outcomes (such as functional capacity, health status, quality of life, self-management, psychosocial health, physical activity and self-efficacy) between those who receive dRPM and BEPR+ (dRPM+) vs. those who receive BEPR+ alone.

DETAILED DESCRIPTION:
Background Chronic obstructive pulmonary disease (COPD) represents a major challenge to health and well-being, necessitating the development of effective management strategies. Pulmonary rehabilitation (PR) has emerged as a crucial approach. However, due to the complexity of COPD and the presence of comorbidities, there is a need for an advanced PR program that can address the diverse needs of patients, including better self-management. In response to this challenge, clinicians and researchers at the G.F. MacDonald Centre for Lung Health have created BEPR+. This program addresses the needs of comorbid COPD patients via a more comprehensive comorbidities assessment, collaborative goal setting process to adopt healthier lifestyle behaviors (with a strong emphasize in physical activity), and a protocolized referral process to facilitate a more comprehensive care approach.

A proposed solution to address better patient self-management following PR involves integrating digital remote patient monitoring (dRPM) into BEPR+ (dRPM+), effectively bridging the gap between self-care and healthcare. The dRPM system will collect and transmit patient-generated data to healthcare providers, enabling timely detection of exacerbations and ultimately reducing hospitalizations. Participants will be educated on monitoring trends in their daily vital signs, allowing early identification of abnormalities that may correlate with changes in symptoms and general health status.

Primary Objective: To assess the feasibility and acceptability of the dRPM+ intervention in individuals undergoing PR. More specifically, the primary objectives are as follows:

1. To assess adherence to and completion of the intervention (i.e., do participants complete the PR classes and take daily physiological readings as prescribed?).
2. To assess recruitment and retention rates.
3. To assess the acceptability of the intervention to individuals undergoing PR.
4. To assess the impact on staff workflow and program resources.

Secondary Objectives: To estimate the impact of the program on self-management, self-efficacy, and standard PR outcomes (i.e., functional capacity, health status, general quality of life, psychosocial health, and physical activity) by generating preliminary estimates of the mean difference between groups over time for each outcome measure.

Study design: A randomized parallel-controlled trial will be implemented at the G.F. MacDonald Centre for Lung Health where entire PR classes I(i.e., delivered Tuesday/Thursday or Monday/Wednesday/Friday) will be block randomized according to a random numbers table to receive the intervention (dRPM+) or the control (BEPR+). Both groups will complete survey and questionnaire data at baseline, post-program, and 12-week follow-up using a REDcap database.

Study design A randomized parallel-controlled trial will be implemented at the G.F. MacDonald Centre for Lung Health. Entire PR classes I(i.e., delivered Tuesday/Thursday for 8 weeks or Monday/Wednesday/Friday for 6 weeks.) will be block randomized according to a random numbers table to receive dRPM+ or BEPR+. In addition to the BEPR+ program, both groups will complete survey and questionnaire data at baseline, specific points throughout the program, post-program, and 12-week follow-up using a REDcap database.

Data Analysis: Data will be presented descriptively and encompass all key relevant summary statistics (such as mean, median, standard deviation, and range). These data will cover various aspects, including participant characteristics, the primary feasibility outcome (dRPM data collection rate), study recruitment and retention, program attendance, patient satisfaction, staff time, questionnaire completion rate and time required. Regression analyses will explore changes in the secondary outcomes while controlling for the effects of potential covariates, including age, sex, disease severity, comorbidities and physical activity.

Data Handling and Record Keeping: Data will be stored in a central Redcap database. Patients will all have a unique study code number, the unique identifier in the Redcap database. A comparison of participants who consented, those who declined to join the trial, and those who completed or dropped out of the program will be conducted using student t-tests. The occurrence of adverse events, relevant staffing time, and resource details will be reported as counts along with qualitative descriptions.

ELIGIBILITY:
Inclusion Criteria:

* patients must be enrolled into pulmonary rehabilitation at the G.F. MacDonald Centre for Lung Health with a diagnosis of chronic lung disease (COPD confirmed by post-bronchodilator forced expiratory volume in 1 second by forced vital capacity (FEV1/FVC) ratio of less than 0.7).

Patients must be able to read and communicate in English and willing and able to use digital devices.

Exclusion Criteria:

* Patients with cognitive impairments who are unable to accurately complete questionnaires will also be excluded.
* As part of standard rehabilitation referral procedures, all patients must be ambulatory and not have unstable cardiovascular disease.

Ages: 30 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2023-09-28 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of recruitment and participant retention | 18 months
  A measure of the recruitment and retention of study participants
Adherence | 18 months
  adherence to vital sign monitoring during the 6 or 8 week pulmonary rehabilitation trial and the 12 week follow-up period.
Acceptability | 18 months
  Using a fit for purpose questionnaire to evaluate participant acceptance of the remote patient monitoring system.

SECONDARY OUTCOMES:
Staffing time and resources | 18 months
  An assessment of the time requirement to monitor and respond to remote patient monitoring notifications
Self-efficacy for managing chronic disease-6 items | Baseline, post-program, and 12-week follow-up
  A generic 6-item tool used to measure of patient's confidence in self-managing their chronic health condition(s). Patients are score each item from 0-10,and the average is reported as the score. Higher scores indicate higher self-efficacy.
Partners in Health Self-Management tool | Baseline, post-program, and 12-week follow-up
  A generic self-reported questionnaire used to assess the self-management knowledge and behaviors or people with chronic diseases. Higher scores indicate better self management knowledge and behaviors.
Self-efficacy for exercise and physical activity | Baseline, post-program, and 12-week follow-up
  A nine item self-reported scale describing different situations (weather, boredom, pain, exercising alone, not pleasurable, too busy, feel tired, stress, depressed) that might effect participation in exercise. The scale asks patients to report their confidence to exercise (from 0- not confident to 10-very confident) 3 times a week for 20 minutes each time despite the above situations.
Physical activity levels | Baseline, post-program, and 12-week follow-up
  Using the Fitbit Versa 4 and measuring step count, active minutes, and sleep
Functional exercise capacity assessed by the 6-minute walk test | Baseline, post-program, and 12-week follow-up
  A self-paced standardized walking test with the primary outcome of 6-minute walk distance as proxy for patients' exercise capacity
Health status as assessed by the COPD Assessment Tool | Baseline, post-program, and 12-week follow-up
  A unidimensional 8-items questionnaire to evaluate the impact of symptoms on patients' health status. Higher scores indicate higher degree of symptoms and a poorer health status.
General health related quality of life as assessed by the EuroQol 5 dimensions 5 level (EQ5D5L) questionnaire. | Baseline, post-program, and 12-week follow-up
  A unidimensional tool that assessed the impact of disease on 5 areas of general health

CONTACTS AND LOCATIONS:
Overall Officials: Michael K Stickland, PhD, Principal Investigator — University of Alberta
Locations (1):
- G. F. MacDonald Centre for Lung Health, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No